CLINICAL TRIAL: NCT04917471
Title: The Effect of Dietary Nitrate Supplementation on Red Blood Cell Function in Patients with Type 2 Diabetes
Brief Title: Effect of Nitrate on Red Blood Cell Function in Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, John Pernow, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: NOBLE-DM
Record Dates: First submitted 2021-05-25; First posted 2021-06-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrate-rich beet root juice (Active Comparator): Nitrate-rich Beet root juice 70 ml bid
  Interventions: Dietary Supplement: Beet root juice
- Placebo (Placebo Comparator): Nitrate-depleted beet root juice 70 ml bid
  Interventions: Dietary Supplement: Placebo juice

INTERVENTIONS:
Dietary Supplement: Beet root juice — 70 ml bid
  Arms: Nitrate-rich beet root juice
Dietary Supplement: Placebo juice — 70 ml bid
  Arms: Placebo

SUMMARY:
To investigate the effect of nitrate supplementation on red blood cell function in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes

Exclusion Criteria:

Acute coronary syndrome Vegetarian diet Impaired renal function Absolute indication for proton pump inhibitor Ongoing treatment with organic nitrate Heart failure (ejection fraction <35%) Any condition that interferes with the possibility to fulfill the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage recovery of left ventricular function | 1 week
  Red blood cells are administered to an isolated rodent heart subjected to 25 min global ischemia and 60 min reperfusion. The percentage recovery during reperfusion is determined.

CONTACTS AND LOCATIONS:
Overall Officials: John Pernow, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No